CLINICAL TRIAL: NCT03742778
Title: Incentivizing Reflection and Output in Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 827107-1257
Record Dates: First submitted 2018-11-13; First posted 2018-11-15 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Healthy
Keywords: exercise; Incentives; reflection; output
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incentivizing reflection (Experimental): Participants will receive three texts each week asking a question to reflect on their latest workout, and will receive 500 points for each text they answer. These bonus points are on top of points participants receive for each workout (200 points per workout). Example text: "Which best describes how you felt right after your last workout? 1-Energized, 2-Proud, or 3-Tired? Send your personal reply (e.g., "1")"
  Interventions: Behavioral: Incentivizing reflection
- Incentivizing Exercise (Experimental): Participants will receive three texts each week asking a question for them to reflect on. Regardless of whether or not they respond to the texts, participants receive 500 bonus points for their first three workouts during the week. These bonus points are on top of points participants receive for each workout (200 points per workout). Example text: "Which best describes how you are feeling now? 1-Energized, 2-Proud, or 3-Tired? Send your personal reply (e.g., "1")"
  Interventions: Behavioral: Incentivizing exercise

INTERVENTIONS:
Behavioral: Incentivizing reflection — Participants receive bonus incentives for reflecting on their workouts
  Arms: Incentivizing reflection
Behavioral: Incentivizing exercise — Participants receive bonus incentives for exercising
  Arms: Incentivizing Exercise

SUMMARY:
This study will test whether incentivizing post-workout activities (i.e., reflecting on workouts) is more effective than incentivizing actual workouts. This study has two conditions: reflection condition (with incentives for reflecting on workouts) vs. output (with incentives for working out). The focus of the incentives will be reinforced by three text messages per week and weekly emails.

DETAILED DESCRIPTION:
Gym members register online to participate in a 28-day workout program. Upon registration, participants are assigned to one of two conditions (a condition that incentivizes reflecting on workouts or a condition that incentivizes workouts). Upon registration, participants are prompted to create a workout schedule and are given advice that reflecting on workouts can help build exercise habits. Over the 28-day intervention period, participants receive text message reminders prior to their scheduled workouts and emails reminding them of their schedules. In both conditions, participants receive points every day that they go to the gym, which can be redeemed for a gift card after the intervention period. In the reflection condition, participants can receive bonus points for responding to each of three text messages each week asking about them to reflect on their gym visits. In the output condition, participants receive the same text messages, but receive bonus points for their first three workouts each week, rather than for responding to text messages.

ELIGIBILITY:
Inclusion Criteria:

* 24 Hour Fitness member

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Gym visits per week | During the 28-day intervention period
  Number of days the participant goes to the gym
Gym visits per week | During the 4-week post-intervention period
  Number of days the participant goes to the gym
Gym visits per week | During the 10-week post-intervention period
  Number of days the participant goes to the gym
Whether or not a participant visits the gym in a given week | During the 28-day intervention period
  Binary variable capturing whether or not a participant had any gym visits in a given week
Whether or not a participant visits the gym in a given week | During the 4-week post-intervention period
  Binary variable capturing whether or not a participant had any gym visits in a given week
Whether or not a participant visits the gym in a given week | During the 10-week post-intervention period
  Binary variable capturing whether or not a participant had any gym visits in a given week

SECONDARY OUTCOMES:
Gym visits per week | During the 52-week post-intervention period
  Number of days the participant goes to the gym
Whether or not a participant visits the gym in a given week | During the 52-week post-intervention period
  Binary variable capturing whether or not a participant had any gym visits in a given week

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No